CLINICAL TRIAL: NCT03619759
Title: The Effect of Sugammadex on the Outcome After Colorectal Cancer Surgery
Acronym: Sugammadex
Status: Completed | Type: Observational
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, In-kyong Yi, Clinical assistant professor, Ajou University School of Medicine
Other Study IDs: AJIRB-MED-MDB-18-36
Record Dates: First submitted 2018-07-10; First posted 2018-08-08 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Outcome, Fatal
Keywords: Sugammadex; Colorectal surgery; postoperative complication
MeSH Terms: conditions — Postoperative Complications | interventions — Sugammadex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sugammadex: Patients who used sugammadex Sugammadex 1 vial (200mg) intravenous, at the end surgery, before extubation
  Interventions: Drug: Sugammadex
- Non-sugammadex: Patients who didn't use sugammadex Pyridostigmine 15~20mg intravenous, at the end of surgery, before extubation

INTERVENTIONS:
Drug: Sugammadex — Sugammadex injection as a reverse agent of neuromuscular blocking
  Other Names: Bridion
  Groups: Sugammadex

SUMMARY:
This study is retrospective study. The purpose of this study is checking the effect of sugammadex on the outcome after colorectal surgery. The outcome is compared among the 2 groups, sugammadex group and non-sugammadex group. The primary parameters of outcome are length of stay, readmission rate, postoperative complications, time interval for first successful oral intake.

DETAILED DESCRIPTION:
Abdominal surgery, like colorectal surgery, needs more than moderate neuromuscular block during surgery. After the surgery, reversal agent of neuromuscular blocking agent is given almost every pateints who underwent general anesthesia.

Classic reversal agent is cholinesterase inhibitor, like pyridostigmine and neostigmine. Its action mechanism is competetive antagonist of rocuronium. But cholinesterase inhibitor cannot make complete reversal in moderate or deep neuromuscular block. Its incomplete reversal which is called residual block cause respiratory complications and prolongation hospital stay.

Sugammadex has different mechanism compared to cholinesterase inhibitor. It captures neuromuscular agent, especially rocuronium, and prevent rocuronium's action. Even in deep neuromuscular block, sugammadex can reverse the action of rocuronium, and its reversal effect is fater and more reliable compared to cholinesterase inhibitor.

Previous studies focused on only short term outcome of sugammadex, like postanesthetic care unit (PACU) discharge time, respiratory complications in PACU.

But in this study, longer term outcome will be comapred between sugammadex group and cholinesterase inhibitor group (pyridostigmine).

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 21~80
* Subjects who took colorectal surgery due to colon or rectal cancer from Jan, 2012 to Dec, 2017

Exclusion criteria

* Emergency surgery
* Paraplegia or quadriplegia
* Bedridden state d/t various reason
* Neuromuscular disease
* Combined operation wth other surgery

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 21 and 80 years old, who took the colorectal surgery due to colorectal cancer from Jan, 2012 to Dec, 2017
Sampling Method: Non-Probability Sample
Enrollment: 585 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Length of stay | admission to discharge (within 1 month)
  Length of stay in hospital

SECONDARY OUTCOMES:
Readmission rate | 30 days after discharge
  Readmission or ER visit within 30 days after discharge
postoperative complication rate | after colorectal surgery, within 30 days
  postoperative complications, heart, lung, kidney, neurovascular, infection etc Check by review discharge summary note, consultation note, and postoperative laboratory tests
Time to first successful oral intake | within 30 days
  time interval between end of surgery and the first successful oral intake

CONTACTS AND LOCATIONS:
Overall Officials: In Kyong Yi, MD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou university school of medicine, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No
No sharing